CLINICAL TRIAL: NCT04954027
Title: Place of Attachment as a Post-weaning Prognostic Factor: Interest of the Implicit Approach
Brief Title: Attachment and Prognostic Factor: the Implicit Approach
Acronym: AIA
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00432-39
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Dependence Addictive
Keywords: implicit approach; post-weaning prognostic factor
MeSH Terms: conditions — Behavior, Addictive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a use-related disorder weaning for a substance
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — 5 visits are planned during the study :
  * the inclusion visit : during this visit the patient's non-opposition is obtained and then the patient answer to self-administered questionnaires online
  * 4 telephone interviews for follow-up by investigator

SUMMARY:
This is a prospective longitudinal study aimed at better understanding the determinants of the prognosis of patients with substance dependence.

5 visits are planned during the study :

* the inclusion visit : during this visit the patient's non-opposition is obtained and then the patient answer to self-administered questionnaires online
* 4 telephone interviews for follow-up by investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years old
* Patients with a use-related disorder as defined by DSM5
* Patients weaning for a substance, supported within the addictology sector of Henri Laborit Hospital
* Having expressed non-opposition to participating in the study after receiving written information.

Exclusion Criteria:

* Person who cannot read or write
* Simultaneous participation in a therapeutic trial involving oxytocin
* Patients protected by law
* Patients who do not have French as their native language
* Patients who, in the opinion of the investigator, are unable to complete the questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a use-related disorder weaning for a substance, supported within the addictology sector of Henri Laborit Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Implicit attachment and onsumption | 12 months
  Assessment of the link between implicit attachment and changes in consumption after a 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried SERRA, Dr, Principal Investigator — Centre Hospitalier Henri Laborit

IPD SHARING:
Plan to Share IPD: No